CLINICAL TRIAL: NCT04896606
Title: A Pilot Study of SARS-CoV-2 Specific Cytotoxic T Lymphocytes (SARS-CoV-2-CTLs) for Treatment of Mild to Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: SARS-CoV-2 CTLS for Mild to Moderate COVID-19 Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Medical College of Wisconsin (Other); Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 604
Record Dates: First submitted 2021-05-19; First posted 2021-05-21 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A run-in pilot will be done treating patients with COVID CTLs for safety. If there are no DLTs per definition in the study, study will proceed with a randomized trial of COVID CTLs + standard of care versus just standard of care alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SARS-CoV-2 CTLS + Standard of Care (Experimental): Patients will get family donor derived SARS-CoV-2 cytotoxic t-lymphocytes up to 5 times every 2 weeks along with Standard of care of COVID-19.
  Interventions: Other: Standard of Care; Biological: SARS-CoV2-CTLS
- Standard of Care Only (Active Comparator): Patients will NOT received COVID CTLs but will get standard of care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Patients will receive standard of care for COVID-19.
Biological: SARS-CoV2-CTLS — Patients may receive up to 5 CTL infusions to treat SARA-CoV-2 in combination with standard of care.
  Arms: SARS-CoV-2 CTLS + Standard of Care

SUMMARY:
The 2019 Severe Acute Respiratory Syndrome (SARS) is a global pandemic secondary to a novel coronavirus - SARS-CoV-2. The reported case-fatality ratio for SARS-CoV-2 in the United States is 1.8% with a current death toll of >300,000 and climbing.4 There is no accepted standard of care or FDA approved therapies for treatment of COVID-19. Virus specific cytotoxic T lymphocytes (CTLs) have become an important part of the treatment landscape for viral reactivation post hematopoietic and solid organ transplantation. Donor derived CTLs have been shown to be safe and effective against a variety of viruses including CMV, EBV, BK and adenovirus. We hypothesize that SARS-CoV-2 specific CTLs generated from a previously infected family donor will be safe and effective for treatment of COVID-19 in family members with mild to moderate disease.

ELIGIBILITY:
INCLUSION CRITERIA

* Age ≥18 to 65 years. AND
* Proven infection with SARS-CoV-2, defined as detection of SARS-CoV-2 by RT-PCR from nasopharyngeal swab or lower respiratory tract specimen AND
* Hospitalized at the time of enrollment AND
* HLA Matched Family Related donor with recent SARS-CoV-2 infection is at least 10 days out from symptom onset. A negative result for COVID-19 by a diagnostic test is not necessary to qualify the donor AND
* In Stage I or II of disease (mild or moderate) at the time of enrollment (Table 1) AND
* ONE of the following high-risk conditions:

  * Chronic lung disease not requiring oxygen at home prior to admission (including but not limited to COPD, cystic fibrosis, asthma and sickle cell disease); Underlying heart disease (including hypertension); Patients with an acute myocardial infarction within the last 3 months will require cardiology clearance prior to enrollment; Diabetes mellitus (type I or II) ; Obesity (BMI ≥ 30); Immunosuppressed, based on investigator's assessment.

EXCLUSION CRITERIA:

* Stage III disease (severe) at the time of enrollment (see Table 1)
* Lack of an identified eligible HLA family related donor
* No high-risk comorbidities defined in the inclusion criteria (Section 5.1)
* Patient with acute GVHD > grade 2 or extensive chronic GVHD at the time of enrollment
* Patient treated with donor lymphocyte infusion (DLI) within 4 weeks prior to CTL Infusion
* Patients with chronic respiratory failure requiring ventilator support and/or oxygen at home prior to admission are excluded
* Patients with stage D heart failure and/or symptoms at rest are excluded
* Renal function: patients with eGFR or CrCl <30 mL/min/1.73 m2 will be excluded from study entry.
* Liver function: Total bilirubin > 2 mg/dl (unless Gilbert's syndrome) OR ALT/AST > 5 x ULN
* Patients currently listed for transplant or potentially eligible to receive organ transplants are excluded from this study
* Patient with poor performance status determined by Karnofsky (patients >16 years) or Lansky (patients ≤16 years) score ≤50%
* Female patient of childbearing age who is pregnant or breast-feeding or not willing to use an effective method of birth control during study treatment and for at least 6 weeks after the last dose of SARS-CoV-2 CTLS.
* Male subjects with female partners of childbearing age who are not willing to use an effective method of birth control during study treatment and for at least 6 weeks after the last dose of SARS-CoV-2 CTLS.
* Concurrent use of following medications is prohibited:

  * Steroids (>2 mg/kg/day prednisone equivalent); Immunotherapies within 4 weeks prior to CTL infusion including checkpoint blockade, ATG, Campath, CAR T cells, blinatumomab; Chemotherapy: Tyrosine kinase inhibitors and hydroxyurea must be stopped > 72 hours prior to SARS-COV-2-CTL cell infusion; High dose chemotherapy must be stopped > 2 weeks prior to SARS-CoV-2-CTLs. High dose chemotherapy is defined in this protocol as any cancer directed therapy causing myelosuppression; Pegylated-asparaginase must be stopped > 4 weeks prior to SARS-COV-2-CTL infusion; Intrathecal chemotherapy must be stopped > 1 week prior to SARS-COV-2-CTL infusion (e.g. intrathecal methotrexate); Anti T-cell Antibodies: Administration of any T cell lytic or toxic antibody (e.g. alemtuzumab) within 30 days prior to SARS-CoV-2-CTLs is prohibited.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 weeks
  no adverse events will occur due to CTL infusion(s)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Study Chair — New York Medical College
Locations (4):
- United States (4):
  - New York Medical College, Valhalla, New York
  - Nationwide Children's Hosptial, Columbus, Ohio
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chu Y, Milner J, Lamb M, Maryamchik E, Rigot O, Ayello J, Harrison L, Shaw R, Behbehani GK, Mardis ER, Miller K, Prakruthi Rao Venkata L, Chang H, Lee D, Rosenthal E, Kadauke S, Bunin N, Talano JA, Johnson B, Wang Y, Cairo MS. Manufacture and Characterization of Good Manufacturing Practice-Compliant SARS-COV-2 Cytotoxic T Lymphocytes. J Infect Dis. 2023 Mar 28;227(6):788-799. doi: 10.1093/infdis/jiac500. PMID 36583990